CLINICAL TRIAL: NCT04588168
Title: Multi-parameter Magnetic Resonance Imaging for Early Evaluation of the Efficacy of Neoadjuvant Chemotherapy With Modified GC Regimen for Urothelial Carcinoma
Brief Title: Multi-parameter Magnetic Resonance Imaging Guides Precise Treatment of Urothelial Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-SR-252
Record Dates: First submitted 2020-09-13; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-09

CONDITIONS: Bladder Cancer
Keywords: Multiparametric Magnetic Resonance Imaging; Bladder Cancer; Chemotherapy
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Drug Therapy; Neoadjuvant Therapy; Cystectomy; Lymph Node Excision; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Chemotherapy + mpMRI + surgery (Experimental): Baseline mpMRI /Neoadjuvant chemotherapy /Immediate mpMRI /Cystectomy and Lymphadenectomy / Postoperative pathology
  Drug: Chemotherapy Procedure: Immediate Multiparametric MRI Procedure: Cystectomy and Lymphadenectomy
  Interventions: Drug: Chemotherapy; Diagnostic Test: Immediate Multiparametric MRI; Procedure: Cystectomy and Lymphadenectomy; Diagnostic Test: conventional Multiparametric MRI; Diagnostic Test: Baseline Multiparametric MRI
- Experimental: Chemotherapy + surgery (Experimental): Baseline mpMRI /Neoadjuvant chemotherapy /Cystectomy and Lymphadenectomy / Postoperative pathology
  Drug: Chemotherapy Procedure: Cystectomy and Lymphadenectomy
  Interventions: Drug: Chemotherapy; Procedure: Cystectomy and Lymphadenectomy; Diagnostic Test: conventional Multiparametric MRI; Diagnostic Test: Baseline Multiparametric MRI

INTERVENTIONS:
Drug: Chemotherapy — Patients with muscle invasive bladder cancer will receive modified gemcitabine-cisplatin neoadjuvant chemotherapy prior to radical cystectomy for a period of two months (three 21 day cycles) as part of standard clinical routine.
  Other Names: Neoadjuvant chemotherapy
Diagnostic Test: Immediate Multiparametric MRI — Within 24 hours after the use of cisplatin during the first course of modified GC neoadjuvant chemotherapy, patient considered muscle invasive bladder cancer with baseline mpMRI will receive an immediate mpMRI scan.
  Other Names: Multiparameter magnetic resonance imaging
  Arms: Experimental: Chemotherapy + mpMRI + surgery
Procedure: Cystectomy and Lymphadenectomy — The patient with muscle invasive bladder cancer will undergo radical cystectomy and pelvic lymph node dissection followed by a urinary tract reconstruction.
  Other Names: surgery
Diagnostic Test: conventional Multiparametric MRI — After two and three course of neoadjuvant chemotherapy, patient considered muscle invasive bladder cancer with baseline mpMRI will receive a conventional mpMRI scan.
  Other Names: Multiparameter magnetic resonance imaging
Diagnostic Test: Baseline Multiparametric MRI — Patient considered muscle invasive bladder cancer will receive a baseline mpMRI scan within one week before neoadjuvant chemotherapy.
  Other Names: Multiparameter magnetic resonance imaging

SUMMARY:
Purpose：To evaluate whether immediate multiparametric MRI evaluate the sensitivity of modified neoadjuvant chemotherapy early in patient with muscle invasive bladder cancer（MIBC）.

Rationale：Multiparametric MRI may help detect the early changes of bladder cancer receiving neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
Objective

Primary: To evaluate whether multiparametric MRI can determine the sensitivity of modified neoadjuvant chemotherapy early in patient with muscle invasive bladder cancer（MIBC）.

Secondary：To determine whether multiparametric MRI can predict the prognosis of modified neoadjuvant chemotherapy early in patient with muscle invasive bladder cancer.

Patients may receive neoadjuvant chemotherapy (typically three 21-day courses of modified gemcitabine-cisplatin(GC) therapy) followed by radical cystectomy and lymph node dissection.

Patients with primary bladder cancer or recurrence which is confirmed by pathology of previous biopsy or TURBT, undergo a multiparametric MRI(mpMRI) at baseline to stage the primary tumor. The mpMRI includes T2-weighted MRI, diffusion-weighted imaging, and dynamic contrast enhancement, which will be given a five-point VI-RADS（Vesical Imaging-Reporting And Data System） score by two radiologists specialized in urogenital radiology. Patients considered NMIBC（Non-muscle invasive bladder cancer） with mpMRI will be given TURBT, while patients with MIBC（Muscle invasive bladder cancer）will receive radical cystectomy and lymph node dissection after three 21-day courses of modified gemcitabine-cisplatin neoadjuvant chemotherapy. Patients also undergo an immediate mpMRI scan after one, two, and three cycles of neoadjuvant chemotherapy.

Specimens from the radical cystectomy are then examined by the pathology department as standard routine.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed primary or recurrent bladder cancer.
* Planned to undergo transurethral resection of bladder tumor (TURBT) or modified GC regimen neoadjuvant chemotherapy plus radical total cystectomy.
* 18 years old and older.
* Willing to give valid written informed consent.
* No contraindications to the MRI(magnetic resonance imaging) and MRI contrast agent.

Exclusion Criteria:

* Abnormal liver function (1.5 times higher than normal).
* Glomerular filtration rate < 60ml /min·kg.
* Heart failure.
* Acute myocardial infarction.
* Severe heart and lung disease.
* Hypotension and hypoxia.
* Brain metastases, or other known central nervous system metastases.
* A history of severe central nervous system diseases, including unexplained loss of consciousness or transient ischemic attack.
* Known congenital or acquired immunodeficiency, active hepatitis, active tuberculosis and other active infections, etc.
* Pregnant or lactating women.
* Patients participating in other drug trials.
* Patients with poor general condition (eg malnutrition, dehydration). Behavioral status score (ZPS quintile) ≥ 2.
* Patients with previous autoimmune diseases or existing autoimmune diseases. (including controlled or uncontrolled drugs).
* Patients undergoing organ transplantation (transplantation of liver, kidney, heart, lung and other organs) or those who require long-term administration of immunosuppressive agents due to personal conditions.
* Those who are intolerant or allergic to cytotoxic chemotherapeutic drugs.
* Bone marrow transplantation, severe leukopenia.
* Patients with severe infection or trauma.
* Any condition based on the investigation's clinical judgment that the patient is not suitable for completing this study (such as not meeting the patient's most beneficial treatment, patient compliance, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline tumor mp-MRI parameters at immediate mp-MRI evaluation. | baseline, during the intervention (Within 24 hours after use of cisplatin of the first course of neoadjuvant chemotherapy(NAC), up to 2 weeks)
  Using the built-in tools of the MRI imaging system to assess the changes of tumor size between immediate mp-MRI evaluation and baseline mp-MRI evaluation after the use of cisplatin during the first course of modified GC neoadjuvant chemotherapy.

SECONDARY OUTCOMES:
Changes from baseline tumor mp-MRI parameters after two course of modified GC neoadjuvant chemotherapy. | baseline, during the intervention(From the end date of the second course of NAC until one day before the third course of NAC, up to 7 weeks)
  Using the built-in tools of the MRI imaging system to assess the changes of tumor size conventional mp-MRI evaluation and baseline mp-MRI evaluation after the second course of modified GC neoadjuvant chemotherapy.
Changes from baseline tumor mp-MRI parameters after three course of modified GC neoadjuvant chemotherapy. | baseline, during the intervention(From the end date of the third course of NAC until one day before surgery, up to 10 weeks)
  Using the built-in tools of the MRI imaging system to assess the changes of tumor size between conventional mp-MRI evaluation and baseline mp-MRI evaluation after the third course of modified GC neoadjuvant chemotherapy.

OTHER OUTCOMES:
Overall survival. | through study completion，an average of 3 year
  Evaluate the overall survival of patients accept the modified GC neoadjuvant chemotherapy followed by radical cystectomy and lymphadenectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Lv Qiang, MD，PHD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first affiliated hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raghavan D. Chemotherapy and cystectomy for invasive transitional cell carcinoma of bladder. Urol Oncol. 2003 Nov-Dec;21(6):468-74. doi: 10.1016/s1078-1439(03)00145-5. PMID 14693275
- [Background] Stein JP, Lieskovsky G, Cote R, Groshen S, Feng AC, Boyd S, Skinner E, Bochner B, Thangathurai D, Mikhail M, Raghavan D, Skinner DG. Radical cystectomy in the treatment of invasive bladder cancer: long-term results in 1,054 patients. J Clin Oncol. 2001 Feb 1;19(3):666-75. doi: 10.1200/JCO.2001.19.3.666. PMID 11157016
- [Background] Grossman HB, Natale RB, Tangen CM, Speights VO, Vogelzang NJ, Trump DL, deVere White RW, Sarosdy MF, Wood DP Jr, Raghavan D, Crawford ED. Neoadjuvant chemotherapy plus cystectomy compared with cystectomy alone for locally advanced bladder cancer. N Engl J Med. 2003 Aug 28;349(9):859-66. doi: 10.1056/NEJMoa022148. PMID 12944571
- [Background] Galsky MD, Pal SK, Chowdhury S, Harshman LC, Crabb SJ, Wong YN, Yu EY, Powles T, Moshier EL, Ladoire S, Hussain SA, Agarwal N, Vaishampayan UN, Recine F, Berthold D, Necchi A, Theodore C, Milowsky MI, Bellmunt J, Rosenberg JE; Retrospective International Study of Cancers of the Urothelial Tract (RISC) Investigators. Comparative effectiveness of gemcitabine plus cisplatin versus methotrexate, vinblastine, doxorubicin, plus cisplatin as neoadjuvant therapy for muscle-invasive bladder cancer. Cancer. 2015 Aug 1;121(15):2586-93. doi: 10.1002/cncr.29387. Epub 2015 Apr 14. PMID 25872978
- [Background] International Collaboration of Trialists; Medical Research Council Advanced Bladder Cancer Working Party (now the National Cancer Research Institute Bladder Cancer Clinical Studies Group); European Organisation for Research and Treatment of Cancer Genito-Urinary Tract Cancer Group; Australian Bladder Cancer Study Group; National Cancer Institute of Canada Clinical Trials Group; Finnbladder; Norwegian Bladder Cancer Study Group; Club Urologico Espanol de Tratamiento Oncologico Group; Griffiths G, Hall R, Sylvester R, Raghavan D, Parmar MK. International phase III trial assessing neoadjuvant cisplatin, methotrexate, and vinblastine chemotherapy for muscle-invasive bladder cancer: long-term results of the BA06 30894 trial. J Clin Oncol. 2011 Jun 1;29(16):2171-7. doi: 10.1200/JCO.2010.32.3139. Epub 2011 Apr 18. PMID 21502557
- [Background] Kim TJ, Cho KS, Koo KC. Current Status and Future Perspectives of Immunotherapy for Locally Advanced or Metastatic Urothelial Carcinoma: A Comprehensive Review. Cancers (Basel). 2020 Jan 13;12(1):192. doi: 10.3390/cancers12010192. PMID 31940998
- [Background] Yin M, Joshi M, Meijer RP, Glantz M, Holder S, Harvey HA, Kaag M, Fransen van de Putte EE, Horenblas S, Drabick JJ. Neoadjuvant Chemotherapy for Muscle-Invasive Bladder Cancer: A Systematic Review and Two-Step Meta-Analysis. Oncologist. 2016 Jun;21(6):708-15. doi: 10.1634/theoncologist.2015-0440. Epub 2016 Apr 6. PMID 27053504
- [Background] Bellmunt J, Mottet N, De Santis M. Urothelial carcinoma management in elderly or unfit patients. EJC Suppl. 2016 Mar;14(1):1-20. doi: 10.1016/j.ejcsup.2016.01.001. Epub 2016 Mar 22. No abstract available. PMID 27358584
- [Background] Galsky MD, Hahn NM, Rosenberg J, Sonpavde G, Hutson T, Oh WK, Dreicer R, Vogelzang N, Sternberg C, Bajorin DF, Bellmunt J. A consensus definition of patients with metastatic urothelial carcinoma who are unfit for cisplatin-based chemotherapy. Lancet Oncol. 2011 Mar;12(3):211-4. doi: 10.1016/S1470-2045(10)70275-8. No abstract available. PMID 21376284
- [Background] Dash A, Galsky MD, Vickers AJ, Serio AM, Koppie TM, Dalbagni G, Bochner BH. Impact of renal impairment on eligibility for adjuvant cisplatin-based chemotherapy in patients with urothelial carcinoma of the bladder. Cancer. 2006 Aug 1;107(3):506-13. doi: 10.1002/cncr.22031. PMID 16773629
- [Background] von der Maase H, Sengelov L, Roberts JT, Ricci S, Dogliotti L, Oliver T, Moore MJ, Zimmermann A, Arning M. Long-term survival results of a randomized trial comparing gemcitabine plus cisplatin, with methotrexate, vinblastine, doxorubicin, plus cisplatin in patients with bladder cancer. J Clin Oncol. 2005 Jul 20;23(21):4602-8. doi: 10.1200/JCO.2005.07.757. PMID 16034041
- [Background] Hayashi N, Tochigi H, Shiraishi T, Takeda K, Kawamura J. A new staging criterion for bladder carcinoma using gadolinium-enhanced magnetic resonance imaging with an endorectal surface coil: a comparison with ultrasonography. BJU Int. 2000 Jan;85(1):32-6. doi: 10.1046/j.1464-410x.2000.00358.x. PMID 10619941
- [Background] Panebianco V, Narumi Y, Altun E, Bochner BH, Efstathiou JA, Hafeez S, Huddart R, Kennish S, Lerner S, Montironi R, Muglia VF, Salomon G, Thomas S, Vargas HA, Witjes JA, Takeuchi M, Barentsz J, Catto JWF. Multiparametric Magnetic Resonance Imaging for Bladder Cancer: Development of VI-RADS (Vesical Imaging-Reporting And Data System). Eur Urol. 2018 Sep;74(3):294-306. doi: 10.1016/j.eururo.2018.04.029. Epub 2018 May 10. PMID 29755006
- [Background] Zargar H, Espiritu PN, Fairey AS, Mertens LS, Dinney CP, Mir MC, Krabbe LM, Cookson MS, Jacobsen NE, Gandhi NM, Griffin J, Montgomery JS, Vasdev N, Yu EY, Youssef D, Xylinas E, Campain NJ, Kassouf W, Dall'Era MA, Seah JA, Ercole CE, Horenblas S, Sridhar SS, McGrath JS, Aning J, Shariat SF, Wright JL, Thorpe AC, Morgan TM, Holzbeierlein JM, Bivalacqua TJ, North S, Barocas DA, Lotan Y, Garcia JA, Stephenson AJ, Shah JB, van Rhijn BW, Daneshmand S, Spiess PE, Black PC. Multicenter assessment of neoadjuvant chemotherapy for muscle-invasive bladder cancer. Eur Urol. 2015 Feb;67(2):241-9. doi: 10.1016/j.eururo.2014.09.007. Epub 2014 Sep 23. PMID 25257030